CLINICAL TRIAL: NCT04157270
Title: LOTUS: Global Acute Stroke Study Utilizing Penumbra System
Acronym: LOTUS
Status: Terminated | Type: Observational
Why Stopped: Business decision to focus on other studies. No safety concern
Sponsor: Penumbra Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: CLP 14788
Record Dates: First submitted 2019-10-04; First posted 2019-11-08 (Actual); Last update posted 2021-06-25 (Actual); Status verified 2021-06

CONDITIONS: Stroke, Ischemic
Keywords: Large Vessel Occlusion; LVO; Mechanical Thrombectomy; Penumbra System
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 90 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Patients with acute ischemic stroke: Patients with acute ischemic stroke secondary to intracranial large vessel occlusion (LVO)
  Interventions: Device: Penumbra System

INTERVENTIONS:
Device: Penumbra System — Penumbra System

SUMMARY:
The primary objective of this study is to demonstrate safety and effectiveness of the Penumbra System in a population with acute ischemic stroke (AIS) secondary to intracranial large vessel occlusion (LVO).

ELIGIBILITY:
Inclusion Criteria:

* Patient age ≥ 18 and ≤ 85
* Patient experiencing acute ischemic stroke secondary to intracranial large vessel occlusion who are eligible for mechanical thrombectomy using the Penumbra System
* Planned frontline treatment with aspiration utilizing Penumbra System
* Present with symptoms consistent with an acute ischemic stroke within 8 hours of stroke symptom onset
* National Institute of Health Stroke Scale (NIHSS) ≥ 6
* Signed informed consent per Institution Review Board/Ethics Committee
* CT ASPECT score from 6 to 10 (≥ 6) or according to MR DWI ASPECT score from 5 to 10 (≥ 5)
* Pre-stroke mRS 0-1

Exclusion Criteria:

* Any comorbid disease or condition expected to compromise survival or ability to complete follow-up assessments through 90 days
* Associated myocardial infarction or severe infection (endocarditis or sepsis)
* Laboratory evidence of coagulation abnormalities, with an International Normalized Ratio (INR) or > 3.0 or platelets count < 40 x 10^9/L or PTT/APTT > 50 sec
* Uncontrolled hypertension (defined as systolic blood pressure > 185 mmHg or diastolic blood pressure > 110 mmHg)
* Baseline glucose < 2.7 or > 22.2 mmol/L
* Seizure at the onset of stroke
* Time of stroke symptom onset unknown
* Females who are pregnant
* Known serious sensitivity to radiographic contrast media that cannot be pre-treated
* Renal failure as defined by serum creatinine > 3.0mg/dl (264 µmol/L)
* Currently participating in an investigational (drug, device, etc.) clinical trial that will confound study endpoints. Patients in observational, natural history, and/or epidemiological studies not involving intervention are eligible
* CT/MRI evidence of the following conditions at screening: significant mass effect with midline shift, evidence of intracranial hemorrhage (ICH), aneurysm, or arteriovenous malformation (AVM), or intracranial tumor
* . Angiographic evidence of preexisting arterial injury, such as carotid dissection, complete cervical carotid occlusion, or vasculitis.
* Angiographic evidence of occlusions in multiple vascular territories (e.g., bilateral anterior circulation, or anterior circulation/vertebrobasilar system) as confirmed on CTA/MRA, or clinical evidence of bilateral strokes or strokes in multiple territories
* Excessive arterial tortuosity that would prevent the device from reaching the target vessel

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients experiencing acute ischemic stroke secondary to intracranial large vessel occlusion who are eligible for mechanical thrombectomy using the Penumbra System
Sampling Method: Non-Probability Sample
Enrollment: 23 (Actual)
Dates: Start 2020-01-12 (Actual); Primary Completion 2021-05-10 (Actual); Study Completion 2021-05-10 (Actual)

PRIMARY OUTCOMES:
mTICI Score | Immediate Post Procedure
  Angiographic revascularization of the occluded target vessel at immediate post-procedure as defined by a modified treatment in cerebral infarction (mTICI) score of 2b or higher. mTICI scale ranges from 0 to 3 with higher values representing better outcomes.
Functional Subject Outcome | 90 days post
  Good functional subject outcome at 90 days post-procedure as defined by modified Rankin Scale (mRS) 0-2. mRS scale from from 0 to 6 with higher values representing a worse outcome.
All-cause mortality at 90 days | 90 days
  All-cause mortality at 90 days

SECONDARY OUTCOMES:
Safety: Device and procedure related SAE | Up to 30 days Post Procedure
  Incidence of device and procedure related Serious Adverse Events (SAEs)
Safety: Occurrence of ENT | Immediate Post Procedure
  Occurrence of embolization in previously uninvolved (or new) territories (ENT) as seen on the final control angiogram at the end of procedure
Safety: Occurrence of Symptomatic intracranial hemorrhage | Up to 24 Hours Post Procedure
  Occurrence of symptomatic hemorrhages (sICH) at 24 hours
Procedural Time | Immediate Post Procedure
  Time from the arterial puncture to revascularization defined by mTICI 2b or greater
Stroke Onset to Revascularization | Immediate Post Procedure
  Time from stroke onset to revascularization defined by mTICI 2b or greater
Complete Revascularization | Immediate Post Procedure
  Complete revascularization, defined as mTICI 2c and 3
Length of index hospital stay | Up to 90 days Post Procedure
Type of Discharge Facility | Up to 90 days Post Procedure

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - RIA, Englewood, Colorado
  - Tampa General Hospital/USF, Tampa, Florida

IPD SHARING:
Plan to Share IPD: Undecided